CLINICAL TRIAL: NCT06865989
Title: Safety and Efficacy of the Omnipod® SmartAdjust 2.0 System Compared to the Omnipod® 5 System in Individuals With Type 1 or Type 2 Diabetes
Brief Title: Omnipod® SmartAdjust 2.0 System Compared to the Omnipod® 5 System in Individuals With Type 1 or Type 2 Diabetes
Acronym: STRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STRIVE
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 1, Type 2
Keywords: T1D; Omnipod; Omnipod 5; T2D
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized two-sequence, multi-center crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Omnipod 5 SmartAdjust 2.0 System (Experimental): A subset of participants will begin the study using the Omnipod 5 SmartAdjust 2.0 System then switch to the comparator, and back again to the experimental system.
  Interventions: Device: Omnipod 5 SmartAdjust 2.0 System; Device: Omnipod 5 System
- Omnipod 5 System (Active Comparator): A subset of participants will begin the study using the Omnipod 5 System then switch to the experimental system for the remainder of the study.
  Interventions: Device: Omnipod 5 SmartAdjust 2.0 System; Device: Omnipod 5 System

INTERVENTIONS:
Device: Omnipod 5 SmartAdjust 2.0 System — Omnipod 5 System with changes
Device: Omnipod 5 System — Cleared device as comparator

SUMMARY:
The goal of this multi-center, randomized, cross-over study is to evaluate the safety and effectiveness of the Omnipod 5 SmartAdjust 2.0 System in individuals with type 1 or type 2 diabetes.

Study participants will complete about 5 in-person visits and be expected to treat their diabetes per their usual routine using the system at the lowest available target setting.

Each participant will begin the study using either the Omnipod 5 SmartAdjust 2.0 System or the Omnipod 5 System for 4 weeks (Period 1) then switch to the opposite system for the next 4 weeks (Period 2). Everyone will use the Omnipod 5 SmartAdjust 2.0 System for the last 4-6 weeks (Period 3). During Period 3, participants will have a goal of administering no more than 3 meal or snack boluses per day.

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of consent 2-70 years (inclusive)
2. Diabetes diagnosis, based on Investigators clinical judgement, and meets the following:

   Diagnosed with type 1 diabetes for at least 3 months for participants aged 2 - < 7 years and at least 1 year for participants aged 7 - 70 years. OR 18-70 years old, diagnosed with type 2 diabetes for at least 1 year
3. Living with a parent or guardian if < 18 years old
4. Omnipod 5 user who has used U-100 insulin or their generic equivalents with the Omnipod 5 system for at least 3 months prior to screening
5. Must have used the target of 110mg/dl for at least 30% of the time for 2-13 year olds and for at least 50% of the time for 14-70 year olds for the 2 weeks preceding the screening visit
6. Willing to use only the following types of U-100 insulin during the study: Humalog U-100, Novolog, or Admelog or their generic equivalents
7. Participant agrees to provide their own insulin for the duration of the study
8. Stable doses over the preceding 4 weeks of non-insulin glucose lowering or weight loss medications that have a meaningful effect on glycemia, as determined by the investigator
9. Investigator has confidence that the participant and/or caregiver can safely operate all study devices and can adhere to the protocol
10. Willing to wear the system continuously throughout the study
11. Willing and able to sign the Informed Consent Form (ICF) or has a parent/guardian willing and able to sign the ICF. Assent will be obtained from pediatric and adolescent participants aged < 18 years per state requirements
12. Able to read and understand English
13. If of childbearing potential, willing and able to have pregnancy testing

Exclusion Criteria:

1. Any medical condition, which in the opinion of the investigator, would put the participant at an unacceptable safety risk
2. Current or known history of coronary artery disease that is not stable with medical management per investigator judgment, including unstable angina, or angina that prevents moderate exercise despite medical management, or a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass grafting within the 12 months prior to screening
3. Any planned surgery during the study which could be considered major in the judgment of the investigator
4. History of severe hypoglycemia in the past 6 months. Severe hypoglycemia is defined as an event that requires the assistance of another person due to altered mental and/or physical status, and requires another person to actively administer carbohydrate, glucagon, or other resuscitative actions.
5. History of diabetic ketoacidosis (DKA) or hyperosmolar hyperglycemic state (HHS) in the past 6 months, unrelated to an intercurrent illness or infusion failure
6. Unable to tolerate adhesive tape or has any unresolved skin condition in the area of sensor or pump placement
7. Blood disorder or dyscrasia within 3 months prior to screening, which in the Investigator's opinion could interfere with determination of HbA1c
8. Use of hydroxyurea
9. Has taken systemic steroids (oral or injectable) within 4 weeks or has had a local steroid injection (e.g. intraarticular, epidural) within 1 week prior to screening or plans to take oral or injectable steroids during the study
10. For type 1 participants only. Use of non-insulin glucose-lowering medication other than metformin and GLP1, in the 4 weeks prior to screening. Participants taking metformin and/or GLP1 should remain on a steady dose during study participation
11. Pregnant or lactating, or of childbearing potential and not on acceptable form of birth control (acceptable forms of contraception include abstinence, barrier methods such as condoms, hormonal contraceptives, intrauterine device, surgical sterilization such as tubal ligation or hysterectomy, or vasectomized partner)
12. In the past 30-days, has participated in a clinical study using any investigational drug or any investigational device. Additionally, may not intend to participate in any other clinical study during this study period.
13. Planned international travel during the study
14. Unable to follow clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the Investigator's clinical judgment
15. Participant is an employee of Insulet, an Investigator or Investigator's study team, or immediate family member of any of the aforementioned

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2025-03-26 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Percent of time in range <54 mg/dL (non-inferiority margin of 0.75%) | End of Period 2 (Day 56) compared to Baseline
  Glucose metric from continuous glucose monitoring system
Percent of time in range <70 mg/dL (non-inferiority margin of 3.0%) | End of Period 2 (Day 56) compared to Baseline
  Glucose metric from continuous glucose monitoring system
Percent of time in range 70-180 mg/dL (non-inferiority margin of 3.0%) | End of Period 2 (Day 56) compared to Baseline
  Glucose metric from continuous glucose monitoring system
Mean Glucose (non-inferiority margin of 8 mg/dL) | End of Period 2 (Day 56) compared to Baseline
  Glucose metric from continuous glucose monitoring system

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Forlenza, MD, Study Chair — Barbara Davis Center
Locations (11):
- United States (11):
  - University of Southern California, Los Angeles, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - Joslin Diabetes Center, Boston, Massachusetts
  - Henry Ford, Detroit, Michigan
  - International Diabetes Center, Minneapolis, Minnesota
  - University Hospitals Cleveland, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas